CLINICAL TRIAL: NCT06218056
Title: Evaluating the Efficacy of Cannabidiol for Reducing Cigarette Use
Brief Title: Cannabidiol for Reducing Cigarette Use
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Edythe London, Distinguished Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-001793
Record Dates: First submitted 2023-12-27; First posted 2024-01-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use Disorder; Tobacco Smoking; Tobacco Dependence
Keywords: Cannabidiol; Tobacco Use Disorder; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Smoking; Smoking Cessation | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (CBD) 800 mg (Active Comparator): Sixty participants who meet all eligibility criteria will be randomized to receive CBD (ATL5; Ananda Scientific) at a dose of 800 mg.
  Interventions: Drug: Cannabidiol (CBD) 800 mg
- Placebo (Placebo Comparator): Sixty participants who meet all eligibility criteria will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol (CBD) 800 mg — CBD (400 mg) will be administered orally twice daily in the morning and again in the evening in 4 capsules each containing 100 mg of the active ingredient in the Ananda investigational new drug, ATL5. ATL5 is cannabidiol (CBD), extracted from hemp, at a 10% strength (softgel capsules with 100 mg/ml of CBD per capsule). The novel formulation is based on the principle that a water-free mixture of some concentrated inactive ingredients (excipients) self-assemble spontaneously into liquid nanodomains that contain the active component CBD. ATL5 Softgel Capsules will be manufactured by Baxco Pharmaceutical Inc., (California, USA) under cGMP conditions.
  Arms: Cannabidiol (CBD) 800 mg
Drug: Placebo — The placebo softgel capsule formulation will have a composition with the same relative proportions as the CBD ATL5 Softgel Capsules. This formulation will be manufactured by Baxco Pharmaceutical Inc under cGMP conditions. 4 softgel capsules of placebo will be administered to match the capsule number of the active compound, daily in the morning and evening for each of 56 days.
  Arms: Placebo

SUMMARY:
The goal of this research is to evaluate the efficacy of cannabidiol (CBD) in reducing cigarette smoking. Although there are safe and effective treatments for smoking cessation, not everyone who attempts smoking cessation is successful, even with these treatments. Relapse rates are high, leaving a need for new approaches. Despite justification to evaluate CBD for this indication, human research on the topic is scant. Larger, more extended studies are warranted and essential.

The investigators will recruit participants from CRI-Help, Inc., a substance abuse treatment program in North Hollywood, where residents who indicate the desire to stop smoking are prohibited from using other cannabis products which would affect recruitment.

The aims of this study are:

1. Evaluate the effects of CBD on changes in cigarette use throughout and following the trial.
2. Exploratory Aims. Measure plasma concentrations of CBD, N-arachidonoyl-ethanolamine (anandamide) and 2-arachidonoylglycerol (2-AG) throughout the trial.

Participants who meet eligibility criteria will take part in a 56-day treatment phase during which they receive the study medication under supervision (CBD or placebo twice daily) and complete questionnaires on side effects, withdrawal, craving and mood symptoms. Blood, breath, and urine tests will also be performed throughout the study. Participants who complete the treatment will also be assessed at 1-month and 3-month follow up visits.

DETAILED DESCRIPTION:
General Experimental Design: This will be a randomized, double-blind, placebo-controlled, comparison study of Nantheia ATL5 (CBD) vs. placebo on smoking behavior in participants who have Tobacco Use Disorder (TUD) and have a desire for smoking cessation, conducted at CRI-Help, Inc., a residential substance use treatment center in N. Hollywood, CA. The investigators will instruct participants and provide support via text messages from the National Cancer Institute's Smokefree.gov website. Smokefree.gov offers free messaging programs that give encouragement, advice, and tips for becoming smoke-free and being healthier. The NCI website also helps people who smoke create a personalized quit plan that makes it easier to stay on track, get through hard times, and quit for good. Creating this plan will be part of baseline procedures.

Randomization to Treatment, Sample Size: Participants will receive CBD at a dose of 800 mg per day or placebo (n = 60/group). The investigators will randomize by sex and age (18-30, greater than/equal to 31 years) to ensure equal representation across the groups. The investigators will use an intention-to-treat analysis, including data from all participants who are randomized (see below for power analysis).

Dosing and Testing Schedule: After screening (Days -7 to 0) and baseline (Day 0) assessments, the study will comprise a 56-day (8-week) treatment period with follow up assessments at 1 and 3 months after termination of treatment as part of this trial. Measurements will be obtained at daily and weekly assessments during the 8-week treatment period.

Measures Collected: A baseline assessment will include assay of blood plasma cotinine to indicate heaviness of smoking, and self-reports of smoking-related behaviors on the following smoking-related questionnaires:

* Fagerström Test for Nicotine Dependence (FTND). This 6-item survey (~2 min) is closely linked to nicotine intake.
* Smoking History Questionnaire. Developed in Dr. London's Lab, this 25-item survey (~5 min) queries age at initiation, longest quit attempt, number of quit attempts, reasons for quitting, and current smoking behavior (e.g., preferred brand, cigarettes per day, etc.).
* Minnesota Nicotine Withdrawal Scale (MNWS) measures withdrawal symptoms: craving, irritability, anxiety, difficulty concentrating, restlessness, headache, drowsiness, and GI disturbances. These symptoms are scored on an ordinal scale [0 (not present) to 3 (severe)].
* General Anxiety Screener (GAD-7). This is a self-administered seven-item questionnaire that is used to measure or assess the severity of generalized anxiety disorder (GAD). The GAD-7 takes ~1-2 min to complete.
* Patient Health Questoinnaire-9 (PHQ-9). This self-administered nine-item scale measures the degree of depression. The PHQ-9 only takes ~1-2 min to complete.

Participants will self-report cigarette use and adverse events (AEs) each day using structured questionnaires. At screening and on days 7, 14, 28 and 56, the investigators will take vital signs and draw blood for clinical laboratory tests for safety, to assay cotinine as an index of heaviness of smoking, and to assay cannabinoids (CBD, anandamide, 2-AG); participants will complete the FTND, MNWS, GAD-7, and PHQ-9. At 1- and 3-month follow up, the investigators will take vital signs, measure CO in breath, and take the same behavioral/self-report measures as on Days 7, 14, 28 and 56.

Retention: The index of retention will be the number of days a participant remains in the study.

Assay of CBD, anandamide, 2-AG and cotinine: The investigators will use liquid chromatography/mass spectrometry-multiple reaction monitoring (LC/MS-MRM) assays. Internal standards are added after sample extracts are processed and injected onto a multi-mode column with reversed phase, cation and anion exchange capabilities. After equilibration and elution, column effluents are passed through an electrospray ion source attached to a triple quadrupole mass spectrometer, and MRM signals are recorded. Each compound is quantified by interpolation from response curves using data from internal standards and increasing concentrations of unlabeled authentic analytes.

Risks and Minimization of Risk

Risks associated with taking CBD include:

* Increase in liver alanine aminotransferase enzymes (ALT test)
* Increase in blood clotting (International Normalized Ratio, INR).

Given the possibility that individuals with substance use disorders will participate in the study and may exhibit abnormality in liver function at baseline, liver function tests will be performed in screening, and individuals with abnormal values will be excluded.

Abuse Potential of CBD: The DEA has classified CBD as a Schedule I drug In the United States, suggesting that CBD has a high potential for abuse, but the World Health Organization Expert Committee on Drug Dependence concluded that no abuse potential could be confirmed based on findings from animal and human research. The type of CBD used here is derived from hemp and contains less than 0.3% tetrahydrocannabinol (THC; i.e., the primary psychoactive ingredient in cannabis). CBD used in Nantheia ATL-5 is not considered a scheduled drug by the DEA.

Note: Careful screening at baseline and ongoing monitoring of plasma levels for potential emergence of adverse events will be practiced, ensuring minimization of all risks.

In addition, trial stopping rules were developed with the following criteria applied.

Patient safety dose stopping and discontinuation criteria (no re-challenge):

* ALT or AST >3 x ULN and [total bilirubin level (TBL) >2 x ULN or INR >1.5).
* ALT or AST >3 x ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (>5%).

Other risks of CBD administration Possible effects on a fetus: There are no long-term studies in humans on CBD effects on fetal development; however, animal studies suggest that long-term use is safe, with very low potential for effects on a fetus at doses associated with human treatment. To minimize this potential risk, pregnancy is an exclusion criterion, and a participant who becomes pregnant will be withdrawn from the study.

Risk of ovarian suppression: Animal studies have indicated this possibility. Female participants will undergo a hormonal battery at screening with ultrasound upon abnormal findings. Participants with evidence of ovarian suppression will be excluded. Ovarian function will also be tested during the treatment phase, and any abnormality followed up with referral for further investigation.

This study will be conducted in a residential treatment facility. Thus, participants will be closely monitored, dosing will be controlled, and clinical and laboratory assessments will be done on a regular schedule.

Participant Withdrawal from the Protocol: Participants can be withdrawn for safety (see stopping criteria above) and noncompliance with medication administration protocols. Decisions regarding safety will be made by the PI with advice from Co-Investigator Larissa Mooney, M.D. Participants will also be withdrawn upon leaving inpatient treatment at CRI-Help. Participants can decide on their own to withdraw from the protocol at any time without prejudice, and this will not affect their treatment at CRI-Help. All participants will receive compensation for all of the procedures/assessments completed.

Drug Administration Details

Investigational Product and Mode of Administration: Nantheia ATL5, which is CBD, extracted from hemp, at a 10% strength (softgel capsules with 100 mg/ml of CBD per capsule) or matching placebo. The formulation that was selected for this clinical trial contains CBD and excipients as here:

1. emulsifying agents: Cremophor EL (Polyoxyl 35 castor oil), Tween 80 (Polysorbate 80), Plurol® Oleique (polyglyceryl-3 dioleate);
2. cwe o-surfactant: propylene glycol;
3. oil: Labrosol® (caprylocapryol polyoxyl-8 glycerides), medium chain triglycerides;
4. antioxidant: BHT (butylated hydroxytoluene).

Nantheia ATL5 Softgel Capsules will be manufactured by Baxco Pharmaceutical Inc. (California, USA), under cGMP conditions for Ananda Therapeutics. Ananda will supply Nantheia ATL5 Softgel Capsules and matching placebo for this study. Capsules will be administered orally as indicated below. Ananda Therapeutics is FDA-approved to supply this product.

Dosage and Duration of Treatment: This study will evaluate Nantheia ATL5 in participants given CBD or placebo (1:1). The treatment period will be 56 days (8 weeks). Participants will be in the study for up to 24 weeks, including follow-up at 1 and 3 months after completion of the treatment protocol. The CBD/placebo dose will be 800 mg/day. Dose Justification: A daily dose of 600 mg is being evaluated in our ongoing trial of CBD for opioid use disorder (ClinicalTrials.gov Identifier: NCT03787628). Doses of CBD as high as 50 mg/kg (i.e., 3500 mg for a 70-kg participant) were well tolerated; and doses between 300 and 1500 mg have been used in humans without serious adverse events. Forty-two subjects received 200 mg of CBD 4x daily (total 800 mg per day) for 2-4 weeks to treat schizophrenia without notable side effects. Additionally, a review of 132 reports including animal and human studies concluded that CBD was well-tolerated in humans, at doses of up to 1500 mg/day.

Regulatory Considerations: CBD will be administered in this protocol as Nantheia ATL5, a hemp-derived product that contains < 0.3% tetrahydrocannabinol (THC). Nantheia ATL5 is not a Schedule 1 controlled substance because Nantheia ATL5 is hemp-derived CBD with a THC concentration of no more than 0.3%. The investigators have obtained FDA approval for this project. The investigators will receive oversight and obtain approval from the UCLA Institutional Review Board.

Receipt and Storage of the Investigational Product (IP). The IP will be delivered by the manufacturer in bottles containing 28 1-mL softgels each for testing of 800 mg CBD vs. placebo. Nantheia ATL5 will be stored at room temperature, 59-86°F (15-30°C), in a locked cabinet in a locked office of a staff member blinded to its identity (CBD or placebo).

Dispensation of the IP: Staff not involved in data entry or any other aspects of the study will distribute the IP into containers labeled with the subject-ID number and/or patient initials and doses will be divided for AM or PM. The investigational product (CBD or placebo) will be taken under staff supervision at the CRI-Help treatment center. A Residential Technician (RADT) will be responsible for supervising and recording patient's self-administration of the IP. Unused or missed medication will be collected once weekly and prepared for return to the manufacturer.

ELIGIBILITY:
Inclusion Criteria:

The investigators will study equal numbers of males and females betweeen 18 - 65 years of age who have Tobacco Use Disorder and express a desire for smoking cessation. Participants will be recruited from the clientele base at Cri-Help Treatment Center in North Hollywood, CA, where the investigators have a long-standing relationship and where the investigators have conducted other research protocols. This study will be conducted at Cri-Help Treatment Center.

Participants will not be recruited from the general population for this study because common use of cannabis in the greater Los Angeles area would confound measurements of CBD, interfering with evaluation of the association of plasma level from treatment with efficacy. This problem is avoided in studying participants who are receiving treatment at a facility where cannabis use is not allowed.

The investigators will include all racial and ethnic groups. Based on the population of the surrounding communities in the Los Angeles region, the investigators anticipate a racial and ethnic makeup of approximately 26% White, 9% Black/African American, 49% Hispanic/Latino, 14% Asian American, and 2% multi-racial/unknown. These percentages align with our recent studies.

Smoking cigarettes and at least moderate nicotine dependence, as indicated by smoking 5 or more cigarettes per day and/or a score of at least 4 on the Fagerström Test for Nicotine Dependence are inclusion criteria. Although vaping is popular and a high proportion of participants who vape also report cigarette smoking (58%), the investigators will exclude participants who vape nicotine. Vaping is not allowed at Cri-Help, Inc.

Exclusion Criteria:

* Physiological dependence on alcohol or any drug, requiring medical detoxification and/or showing signs of acute withdrawal symptoms from opioids, alcohol or benzodiazepines.
* Treatment of Opioid Use Disorder with buprenorphine or methadone to avoid potential drug-drug interactions. CBD interacts with CYP3A. Opioid drugs metabolized by cytochrome P450 (CYP450), and cytochrome P450 isoenzyme CYP3A4 (CYP3A4) in particular, include fentanyl, methadone, oxycodone, and buprenorphine.
* Meeting DSM-5 criteria for schizophrenia, Bipolar I disorder, psychotic disorder, having active suicidal ideation, or suicide attempt in the past 12 months. NOTE: Participants with other psychiatric conditions, such as major depression, generalized anxiety, dysthymia, social phobia or specific phobia can enroll if they are clinically stable.
* AIDS or current HIV medication treatment with antiviral and/or non-antiviral therapy (due to the interaction of CBD with antiviral therapy).
* Clinically significant abnormalities on EKG (such as evidence of arrhythmia or MI).
* Clinically significant cardiovascular, hematologic, hepatic, renal, neurological, or endocrine abnormalities [specific exclusion criteria: AST greater than or equal to 3Xs ULN, Bilirubin greater or equal to 1.5 X ULN, Prothrombin time/International Normalized Ratio (INR) > 1.5.
* Pregnancy and/or lactation. Contraception methods required at time of enrollment, and throughout the duration of the study medication period include abstinence, oral contraceptives, depot contraceptives, condom with spermicide, cervical cap with spermicide, diaphragm with spermicide, intrauterine device, surgical sterilization (e.g. tubal ligation, vasectomy).
* Because of evidence that CBD affects ovarian function in rats, women with values outside the reference ranges on a hormonal battery [estradiol, follicle- stimulating hormone, free thyroxine index, luteinizing hormone, prolactin, total T3 and total T4, thyroid-stimulating hormone], followed by an abnormal ovarian ultrasound finding will be excluded.
* Based on data obtained using Epidiolex® (CBD) oral solution label section 7, "Drug Interactions", the investigators will exclude participants who are taking the following medications: a) strong inducers of CYP3A4 or CYP2C19, which may decrease CBD plasma levels; and b) substrates of UGT1A9, UGT2B7, CYP2B6, CYP2C19 due to the potential of CBD to inhibit enzyme activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effects of CBD on change in cigarette use | 24 weeks
  Change in cigarette use will be indexed by self-reported number of cigarettes/day.
Validate self-reported effects of CBD on change in cigarette use | 24 weeks
  Plasma levels of cotinine (ng/mL) will be measured to validate self-reported tobacco use.

SECONDARY OUTCOMES:
Abstinence from smoking during the last 2 weeks of the trial | 2 weeks (Days 42-56)
  Abstinence from smoking will be indexed categorically by self-report questionnaires.
Confirmation of abstinence from smoking during the last 2 weeks of the trial | 2 weeks (Days 42-56)
  Self-reported abstinence will be confirmed by point of care measurement of expired carbon monoxide (CO, parts per million, ppm).
Validation of abstinence from smoking during the last 2 weeks of the trial | 2 weeks (Days 42-56)
  Abstinence from smoking during the last 2 weeks of the trial will be confirmed biochemically by measure of plasma cotinine (ng/mL).
Change in nicotine dependence | 8 weeks
  Nicotine dependence will be measured weekly on the Fagerström Test for Nicotine Dependence. It contains six items.
  Yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine.
Change in nicotine withdrawal | 8 weeks
  Nicotine withdrawal will be measured weekly measured weekly on the Minnesota Withdrawal Scale, which measures cigarette craving, irritability, anxiety, difficulty concentrating, restlessness, headache, drowsiness, and gastrointestinal tract disturbances. These symptoms are generally scored on an ordinal scale ranging from 0 (not present) to 3 (severe intensity). A summary score is computed.
Changes in mood state - depression | 24 weeks
  Changes in mood state related to depression will be measured weekly and at 1- and 3-month follow ups using the Patient Health Questionnaire-9 (PHQ-9). This questionnaire contains 9 questions, each scored on a scale from 0-3 indicating frequency of the experience in the past week (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day). The scores for each question are added to generate a Total Score. A higher Total Score indicates a more severe depression outcome. Total Scores of 0 = no depression, 1-4 = minimal depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, and 20-27 = severe depression.
Changes in mood state - anxiety | 24 weeks
  Changes in mood state related to anxiety will be measured weekly and at 1- and 3-month follow ups on the Generalized Anxiety Disorder-7 (GAD-7) questionnaire. The GAD-7 contains 7 questions related to having experienced specific symptoms of anxiety over the past week, scored 0-3, with 0 = not at all, 1 = several days, 2 = more than half the days, and 3 = nearly every day. Scores from each question are added to generate a Total Score. A higher Total Score indicates a more severe anxiety outcome, with 0-4 = minimal anxiety, 5-9 = mild anxiety, 10-14 = moderate anxiety, and 15-21 = severe anxiety.

OTHER OUTCOMES:
Plasma concentrations of CBD | 24 weeks
  The primary endpoint will be CBD plasma level (ng/mL) which will be measured at baseline and regularly throughout the trial.
Plasma concentrations of N-arachidonoyl ethanolamine (anandamide) | 24 weeks
  Anandamide (ng/mL) will be measured at baseline and regularly throughout the trial.
Plasma concentrations of 2-arachidonoylglycerol (2-AG) | 24 weeks
  Levels of 2-AG 9ng/mL) will be measured at baseline and regularly throughout the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Edythe D London, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- CRI-Help, Inc., North Hollywood, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and stored biospecimens can be used in additional research to be conducted by study investigators associated with the Center for Medicinal Cannabis Research (CMCR) conducting IRB approved research. Biospecimens and data collected in the course of the study will be banked and may be sent to other research scientists anonymously (without identification). The CMCR leadership will be responsible for deciding how the biospecimens will be used. Information related to the collection, storage, and possible uses of biospecimens has been included in the consent.
Time Frame: Data will be provided to CMCR and CMCR leadership will decide on requests for data from other investigators -- after the study is complete, expected in December 2026.
Access Criteria: Interested investigators would need to contact CMCR, where criteria will be determined.

REFERENCES:
- [Background] Fusar-Poli P, Crippa JA, Bhattacharyya S, Borgwardt SJ, Allen P, Martin-Santos R, Seal M, Surguladze SA, O'Carrol C, Atakan Z, Zuardi AW, McGuire PK. Distinct effects of delta9-tetrahydrocannabinol and cannabidiol on neural activation during emotional processing. Arch Gen Psychiatry. 2009 Jan;66(1):95-105. doi: 10.1001/archgenpsychiatry.2008.519. PMID 19124693
- [Background] Zuardi AW, Morais SL, Guimaraes FS, Mechoulam R. Antipsychotic effect of cannabidiol. J Clin Psychiatry. 1995 Oct;56(10):485-6. No abstract available. PMID 7559378
- [Background] Zuardi AW, Crippa JA, Hallak JE, Moreira FA, Guimaraes FS. Cannabidiol, a Cannabis sativa constituent, as an antipsychotic drug. Braz J Med Biol Res. 2006 Apr;39(4):421-9. doi: 10.1590/s0100-879x2006000400001. Epub 2006 Apr 3. PMID 16612464
- [Background] Zuardi AW, Cosme RA, Graeff FG, Guimaraes FS. Effects of ipsapirone and cannabidiol on human experimental anxiety. J Psychopharmacol. 1993 Jan;7(1 Suppl):82-8. doi: 10.1177/026988119300700112. PMID 22290374
- [Background] Zuardi AW. Cannabidiol: from an inactive cannabinoid to a drug with wide spectrum of action. Braz J Psychiatry. 2008 Sep;30(3):271-80. doi: 10.1590/s1516-44462008000300015. PMID 18833429
- [Background] Wu P, Wilson K, Dimoulas P, Mills EJ. Effectiveness of smoking cessation therapies: a systematic review and meta-analysis. BMC Public Health. 2006 Dec 11;6:300. doi: 10.1186/1471-2458-6-300. PMID 17156479
- [Background] Wheless JW, Dlugos D, Miller I, Oh DA, Parikh N, Phillips S, Renfroe JB, Roberts CM, Saeed I, Sparagana SP, Yu J, Cilio MR; INS011-14-029 Study Investigators. Pharmacokinetics and Tolerability of Multiple Doses of Pharmaceutical-Grade Synthetic Cannabidiol in Pediatric Patients with Treatment-Resistant Epilepsy. CNS Drugs. 2019 Jun;33(6):593-604. doi: 10.1007/s40263-019-00624-4. PMID 31049885
- [Background] Welty TE, Luebke A, Gidal BE. Cannabidiol: promise and pitfalls. Epilepsy Curr. 2014 Sep;14(5):250-2. doi: 10.5698/1535-7597-14.5.250. PMID 25346628
- [Background] Wakeford AGP, Wetzell BB, Pomfrey RL, Clasen MM, Taylor WW, Hempel BJ, Riley AL. The effects of cannabidiol (CBD) on Delta(9)-tetrahydrocannabinol (THC) self-administration in male and female Long-Evans rats. Exp Clin Psychopharmacol. 2017 Aug;25(4):242-248. doi: 10.1037/pha0000135. Epub 2017 Jul 6. PMID 28682102
- [Background] Spanagel R. Cannabinoids and the endocannabinoid system in reward processing and addiction: from mechanisms to interventions . Dialogues Clin Neurosci. 2020 Sep;22(3):241-250. doi: 10.31887/DCNS.2020.22.3/rspanagel. PMID 33162767
- [Background] Smith LC, Tieu L, Suhandynata RT, Boomhower B, Hoffman M, Sepulveda Y, Carrette LLG, Momper JD, Fitzgerald RL, Hanham K, Dowling J, Kallupi M, George O. Cannabidiol reduces withdrawal symptoms in nicotine-dependent rats. Psychopharmacology (Berl). 2021 Aug;238(8):2201-2211. doi: 10.1007/s00213-021-05845-4. Epub 2021 Apr 28. PMID 33909102
- [Background] Scheidweiler KB, Newmeyer MN, Barnes AJ, Huestis MA. Quantification of cannabinoids and their free and glucuronide metabolites in whole blood by disposable pipette extraction and liquid chromatography-tandem mass spectrometry. J Chromatogr A. 2016 Jul 1;1453:34-42. doi: 10.1016/j.chroma.2016.05.024. Epub 2016 May 7. PMID 27236483
- [Background] Sasco AJ, Secretan MB, Straif K. Tobacco smoking and cancer: a brief review of recent epidemiological evidence. Lung Cancer. 2004 Aug;45 Suppl 2:S3-9. doi: 10.1016/j.lungcan.2004.07.998. PMID 15552776
- [Background] Roslawski MJ, Remmel RP, Karanam A, Leppik IE, Marino SE, Birnbaum AK. Simultaneous Quantification of 13 Cannabinoids and Metabolites in Human Plasma by Liquid Chromatography Tandem Mass Spectrometry in Adult Epilepsy Patients. Ther Drug Monit. 2019 Jun;41(3):357-370. doi: 10.1097/FTD.0000000000000583. PMID 30520828
- [Background] Rosen LJ, Galili T, Kott J, Goodman M, Freedman LS. Diminishing benefit of smoking cessation medications during the first year: a meta-analysis of randomized controlled trials. Addiction. 2018 May;113(5):805-816. doi: 10.1111/add.14134. Epub 2018 Jan 29. PMID 29377409
- [Background] Perucca E, Bialer M. Critical Aspects Affecting Cannabidiol Oral Bioavailability and Metabolic Elimination, and Related Clinical Implications. CNS Drugs. 2020 Aug;34(8):795-800. doi: 10.1007/s40263-020-00741-5. PMID 32504461
- [Background] Pertwee RG. The diverse CB1 and CB2 receptor pharmacology of three plant cannabinoids: delta9-tetrahydrocannabinol, cannabidiol and delta9-tetrahydrocannabivarin. Br J Pharmacol. 2008 Jan;153(2):199-215. doi: 10.1038/sj.bjp.0707442. Epub 2007 Sep 10. PMID 17828291
- [Background] Paulus V, Billieux J, Benyamina A, Karila L. Cannabidiol in the context of substance use disorder treatment: A systematic review. Addict Behav. 2022 Sep;132:107360. doi: 10.1016/j.addbeh.2022.107360. Epub 2022 May 7. PMID 35580370
- [Background] Notley C, Gentry S, Livingstone-Banks J, Bauld L, Perera R, Hartmann-Boyce J. Incentives for smoking cessation. Cochrane Database Syst Rev. 2019 Jul 17;7(7):CD004307. doi: 10.1002/14651858.CD004307.pub6. PMID 31313293
- [Background] Morgan CJ, Das RK, Joye A, Curran HV, Kamboj SK. Cannabidiol reduces cigarette consumption in tobacco smokers: preliminary findings. Addict Behav. 2013 Sep;38(9):2433-6. doi: 10.1016/j.addbeh.2013.03.011. Epub 2013 Apr 1. PMID 23685330
- [Background] Mitrirattanakul S, Ramakul N, Guerrero AV, Matsuka Y, Ono T, Iwase H, Mackie K, Faull KF, Spigelman I. Site-specific increases in peripheral cannabinoid receptors and their endogenous ligands in a model of neuropathic pain. Pain. 2006 Dec 15;126(1-3):102-14. doi: 10.1016/j.pain.2006.06.016. Epub 2006 Jul 14. PMID 16844297
- [Background] McPherson SM, Burduli E, Smith CL, Herron J, Oluwoye O, Hirchak K, Orr MF, McDonell MG, Roll JM. A review of contingency management for the treatment of substance-use disorders: adaptation for underserved populations, use of experimental technologies, and personalized optimization strategies. Subst Abuse Rehabil. 2018 Aug 13;9:43-57. doi: 10.2147/SAR.S138439. eCollection 2018. PMID 30147392
- [Background] Maione S, Piscitelli F, Gatta L, Vita D, De Petrocellis L, Palazzo E, de Novellis V, Di Marzo V. Non-psychoactive cannabinoids modulate the descending pathway of antinociception in anaesthetized rats through several mechanisms of action. Br J Pharmacol. 2011 Feb;162(3):584-96. doi: 10.1111/j.1476-5381.2010.01063.x. PMID 20942863
- [Background] Leweke FM, Piomelli D, Pahlisch F, Muhl D, Gerth CW, Hoyer C, Klosterkotter J, Hellmich M, Koethe D. Cannabidiol enhances anandamide signaling and alleviates psychotic symptoms of schizophrenia. Transl Psychiatry. 2012 Mar 20;2(3):e94. doi: 10.1038/tp.2012.15. PMID 22832859
- [Background] Le Foll B, Forget B, Aubin HJ, Goldberg SR. Blocking cannabinoid CB1 receptors for the treatment of nicotine dependence: insights from pre-clinical and clinical studies. Addict Biol. 2008 Jun;13(2):239-52. doi: 10.1111/j.1369-1600.2008.00113.x. PMID 18482433
- [Background] Kendzor DE, Businelle MS, Poonawalla IB, Cuate EL, Kesh A, Rios DM, Ma P, Balis DS. Financial incentives for abstinence among socioeconomically disadvantaged individuals in smoking cessation treatment. Am J Public Health. 2015 Jun;105(6):1198-205. doi: 10.2105/AJPH.2014.302102. Epub 2014 Nov 13. PMID 25393172
- [Background] Kotlinska-Lemieszek A, Klepstad P, Haugen DF. Clinically significant drug-drug interactions involving opioid analgesics used for pain treatment in patients with cancer: a systematic review. Drug Des Devel Ther. 2015 Sep 16;9:5255-67. doi: 10.2147/DDDT.S86983. eCollection 2015. PMID 26396499
- [Background] Kathmann M, Flau K, Redmer A, Trankle C, Schlicker E. Cannabidiol is an allosteric modulator at mu- and delta-opioid receptors. Naunyn Schmiedebergs Arch Pharmacol. 2006 Feb;372(5):354-61. doi: 10.1007/s00210-006-0033-x. Epub 2006 Feb 18. PMID 16489449
- [Background] Karimi-Haghighi S, Razavi Y, Iezzi D, Scheyer AF, Manzoni O, Haghparast A. Cannabidiol and substance use disorder: Dream or reality. Neuropharmacology. 2022 Apr 1;207:108948. doi: 10.1016/j.neuropharm.2022.108948. Epub 2022 Jan 13. PMID 35032495
- [Background] Jordan CJ, Xi ZX. Discovery and development of varenicline for smoking cessation. Expert Opin Drug Discov. 2018 Jul;13(7):671-683. doi: 10.1080/17460441.2018.1458090. Epub 2018 Mar 28. PMID 29587555
- [Background] Hughes JR, Keely J, Naud S. Shape of the relapse curve and long-term abstinence among untreated smokers. Addiction. 2004 Jan;99(1):29-38. doi: 10.1111/j.1360-0443.2004.00540.x. PMID 14678060
- [Background] Hindocha C, Freeman TP, Grabski M, Crudgington H, Davies AC, Stroud JB, Das RK, Lawn W, Morgan CJA, Curran HV. The effects of cannabidiol on impulsivity and memory during abstinence in cigarette dependent smokers. Sci Rep. 2018 May 15;8(1):7568. doi: 10.1038/s41598-018-25846-2. PMID 29765102
- [Background] Hindocha C, Freeman TP, Grabski M, Stroud JB, Crudgington H, Davies AC, Das RK, Lawn W, Morgan CJA, Curran HV. Cannabidiol reverses attentional bias to cigarette cues in a human experimental model of tobacco withdrawal. Addiction. 2018 May 1;113(9):1696-705. doi: 10.1111/add.14243. Online ahead of print. PMID 29714034
- [Background] Halperin AC, McAfee TA, Jack LM, Catz SL, McClure JB, Deprey TM, Richards J, Zbikowski SM, Swan GE. Impact of symptoms experienced by varenicline users on tobacco treatment in a real world setting. J Subst Abuse Treat. 2009 Jun;36(4):428-34. doi: 10.1016/j.jsat.2008.09.001. Epub 2008 Nov 11. PMID 19004600
- [Background] Garcia-Gomez L, Hernandez-Perez A, Noe-Diaz V, Riesco-Miranda JA, Jimenez-Ruiz C. SMOKING CESSATION TREATMENTS: CURRENT PSYCHOLOGICAL AND PHARMACOLOGICAL OPTIONS. Rev Invest Clin. 2019;71(1):7-16. doi: 10.24875/RIC.18002629. PMID 30810545
- [Background] Gamaleddin IH, Trigo JM, Gueye AB, Zvonok A, Makriyannis A, Goldberg SR, Le Foll B. Role of the endogenous cannabinoid system in nicotine addiction: novel insights. Front Psychiatry. 2015 Mar 25;6:41. doi: 10.3389/fpsyt.2015.00041. eCollection 2015. PMID 25859226
- [Background] Elmes MW, Kaczocha M, Berger WT, Leung K, Ralph BP, Wang L, Sweeney JM, Miyauchi JT, Tsirka SE, Ojima I, Deutsch DG. Fatty acid-binding proteins (FABPs) are intracellular carriers for Delta9-tetrahydrocannabinol (THC) and cannabidiol (CBD). J Biol Chem. 2015 Apr 3;290(14):8711-21. doi: 10.1074/jbc.M114.618447. Epub 2015 Feb 9. PMID 25666611
- [Background] Gomez-Coronado N, Walker AJ, Berk M, Dodd S. Current and Emerging Pharmacotherapies for Cessation of Tobacco Smoking. Pharmacotherapy. 2018 Feb;38(2):235-258. doi: 10.1002/phar.2073. Epub 2018 Jan 29. PMID 29250815
- [Background] Dos Santos RG, Hallak JEC, Crippa JAS. Neuropharmacological Effects of the Main Phytocannabinoids: A Narrative Review. Adv Exp Med Biol. 2021;1264:29-45. doi: 10.1007/978-3-030-57369-0_3. PMID 33332002
- [Background] Devinsky O, Marsh E, Friedman D, Thiele E, Laux L, Sullivan J, Miller I, Flamini R, Wilfong A, Filloux F, Wong M, Tilton N, Bruno P, Bluvstein J, Hedlund J, Kamens R, Maclean J, Nangia S, Singhal NS, Wilson CA, Patel A, Cilio MR. Cannabidiol in patients with treatment-resistant epilepsy: an open-label interventional trial. Lancet Neurol. 2016 Mar;15(3):270-8. doi: 10.1016/S1474-4422(15)00379-8. Epub 2015 Dec 24. PMID 26724101
- [Background] Consroe P, Laguna J, Allender J, Snider S, Stern L, Sandyk R, Kennedy K, Schram K. Controlled clinical trial of cannabidiol in Huntington's disease. Pharmacol Biochem Behav. 1991 Nov;40(3):701-8. doi: 10.1016/0091-3057(91)90386-g. PMID 1839644
- [Background] Businelle MS, Kendzor DE, Kesh A, Cuate EL, Poonawalla IB, Reitzel LR, Okuyemi KS, Wetter DW. Small financial incentives increase smoking cessation in homeless smokers: a pilot study. Addict Behav. 2014 Mar;39(3):717-20. doi: 10.1016/j.addbeh.2013.11.017. Epub 2013 Nov 27. PMID 24321696
- [Background] Burggren AC, Shirazi A, Ginder N, London ED. Cannabis effects on brain structure, function, and cognition: considerations for medical uses of cannabis and its derivatives. Am J Drug Alcohol Abuse. 2019;45(6):563-579. doi: 10.1080/00952990.2019.1634086. Epub 2019 Jul 31. PMID 31365275
- [Background] Borgwardt SJ, Allen P, Bhattacharyya S, Fusar-Poli P, Crippa JA, Seal ML, Fraccaro V, Atakan Z, Martin-Santos R, O'Carroll C, Rubia K, McGuire PK. Neural basis of Delta-9-tetrahydrocannabinol and cannabidiol: effects during response inhibition. Biol Psychiatry. 2008 Dec 1;64(11):966-73. doi: 10.1016/j.biopsych.2008.05.011. Epub 2008 Jun 27. PMID 18589404
- [Background] Bergamaschi MM, Queiroz RH, Zuardi AW, Crippa JA. Safety and side effects of cannabidiol, a Cannabis sativa constituent. Curr Drug Saf. 2011 Sep 1;6(4):237-49. doi: 10.2174/157488611798280924. PMID 22129319
- [Background] Baker TB, Piper ME, Smith SS, Bolt DM, Stein JH, Fiore MC. Effects of Combined Varenicline With Nicotine Patch and of Extended Treatment Duration on Smoking Cessation: A Randomized Clinical Trial. JAMA. 2021 Oct 19;326(15):1485-1493. doi: 10.1001/jama.2021.15333. PMID 34665204
- [Background] Ananda Scientific (2021). ATL-5 Investigator's Brochure.